CLINICAL TRIAL: NCT02899169
Title: Treatment of Non-high-risk Acute Promyelocytic Leukemia With Realgar-Indigo Naturalis Formula (RIF) and All-trans Retinoid Acid (ATRA)
Brief Title: Treatment of Non-high-risk Acute Promyelocytic Leukemia (APL) With Realgar-Indigo Naturalis Formula (RIF)
Acronym: APL16
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2016LSL-017
Record Dates: First submitted 2016-09-04; First posted 2016-09-14 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute promyelocytic leukemia; Realgar-Indigo Naturalis Formula; All-trans Retinoic Acid
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin; Arsenic Trioxide; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Realgar-Indigo naturalis formula(RIF) Group (Experimental): Induction therapy: ATO and ATRA, which will maintain until complete hematologic remission. Hydroxyurea should be administrated until WBC count decrease <10x109/L. Consolidation therapy: RIF（60mg/kg/d) and ATRA 4 weeks on and 2 weeks off, until the fusion gene expression is negative. Maintenance therapy: RIF and ATRA 2 weeks on and 2 weeks off for a total of 6 courses.
  Interventions: Drug: Realgar-Indigo naturalis formula; Drug: all-trans retinoic acid; Drug: Hydroxyurea
- Intravenous Arsenic Trioxide(ATO) Group (Active Comparator): Induction therapy: ATO and ATRA, which will maintain until complete hematologic remission. Hydroxyurea should be administrated until WBC count decrease <10x109/L. Consolidation therapy: ATO and ATRA 4 weeks on and 2 weeks off, until the fusion gene expression is negative. Maintenance therapy: ATO and ATRA 2 weeks on and 2 weeks off for a total of 6 courses.
  Interventions: Drug: all-trans retinoic acid; Drug: Arsenic trioxide; Drug: Hydroxyurea

INTERVENTIONS:
Drug: Realgar-Indigo naturalis formula
  Other Names: RIF
  Arms: Oral Realgar-Indigo naturalis formula(RIF) Group
Drug: all-trans retinoic acid
  Other Names: ATRA; Tretinoin
Drug: Arsenic trioxide
  Other Names: ATO; Trisenox (R); As2O3
  Arms: Intravenous Arsenic Trioxide(ATO) Group
Drug: Hydroxyurea

SUMMARY:
The investigators design a multicenter randomized controlled trial to prove that RIF plus ATRA is possibly superior to ATO plus ATRA as consolidation and maintenance treatment for the patients with non-high-risk APL.

DETAILED DESCRIPTION:
Acute promyelocytic leukemia (APL) is a unique subtype of acute myeloid leukemia (AML) which accounts for 10-15% of acute myeloid leukemia. It is characterized by the PML-RARA fusion gene generated by the t(15;17)(q22;q21) chromosomal translocation. The application of ATRA and ATO, make APL from highly fatal to highly curable. APL0406 study proves that ATRA plus arsenic trioxide is at least not inferior and may be superior to ATRA plus chemotherapy in the treatment of patients with non-high-risk APL. Now, the arsenic trioxide has already became the based regimen as targeted first-line treatment without chemotherapy. A study shows that oral RIF plus ATRA is not inferior to intravenous ATO plus ATRA as maintenance treatment of APL. The investigators design a multicenter randomized controlled trial to prove that RIF plus ATRA is possibly superior to ATO plus ATRA as consolidation and maintenance treatment for the patients with non-high-risk APL. Application of oral RIF decrease the total hospitalization days.

ELIGIBILITY:
Inclusion Criteria:

* age 14 to 70 years
* Newly diagnosed APL with t(15;17)(q22;q12)
* Before treatment the Peripheral blood white blood cell count≤10×109/L
* Patients who can complete the entire treatment process
* Patients or their families signed written informed consent

Exclusion Criteria:

* Be allergic to the drug ingredient, the supplementary material or the allergic constitution person
* Cardiac insufficiency, renal insufficiency, significant arrhythmias, EKG abnormalities or other important organ dysfunction
* Combined with other malignant tumors
* Pregnant and lactating women
* Participants in other drug trials in the last 3 months
* Suffering from mental illness or other circumstances which unable to carry out the plan
* Other patients who were not suitable for the study

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | At 2 years

SECONDARY OUTCOMES:
Rate of overall survival (OS) | At 2 years
Event-free survival | From date of randomization until the date of first documented event, assessed up to 36 months
Rate of cumulative incidence of relapse (CIR) | assessed up to 3 years after randomization
Incidence of hematological and non-hematological toxicity | From date of randomization until 2 years
medical expense | From date of randomization until 2 years
Total hospitalization days during therapy | At 2 years from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Huaiyu Wang, Dr., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lo-Coco F, Avvisati G, Vignetti M, Thiede C, Orlando SM, Iacobelli S, Ferrara F, Fazi P, Cicconi L, Di Bona E, Specchia G, Sica S, Divona M, Levis A, Fiedler W, Cerqui E, Breccia M, Fioritoni G, Salih HR, Cazzola M, Melillo L, Carella AM, Brandts CH, Morra E, von Lilienfeld-Toal M, Hertenstein B, Wattad M, Lubbert M, Hanel M, Schmitz N, Link H, Kropp MG, Rambaldi A, La Nasa G, Luppi M, Ciceri F, Finizio O, Venditti A, Fabbiano F, Dohner K, Sauer M, Ganser A, Amadori S, Mandelli F, Dohner H, Ehninger G, Schlenk RF, Platzbecker U; Gruppo Italiano Malattie Ematologiche dell'Adulto; German-Austrian Acute Myeloid Leukemia Study Group; Study Alliance Leukemia. Retinoic acid and arsenic trioxide for acute promyelocytic leukemia. N Engl J Med. 2013 Jul 11;369(2):111-21. doi: 10.1056/NEJMoa1300874. PMID 23841729
- [Result] Zhu HH, Wu DP, Jin J, Li JY, Ma J, Wang JX, Jiang H, Chen SJ, Huang XJ. Oral tetra-arsenic tetra-sulfide formula versus intravenous arsenic trioxide as first-line treatment of acute promyelocytic leukemia: a multicenter randomized controlled trial. J Clin Oncol. 2013 Nov 20;31(33):4215-21. doi: 10.1200/JCO.2013.48.8312. Epub 2013 Oct 14. PMID 24127444
- [Result] Zhu HH, Huang XJ. Oral arsenic and retinoic acid for non-high-risk acute promyelocytic leukemia. N Engl J Med. 2014 Dec 4;371(23):2239-41. doi: 10.1056/NEJMc1412035. No abstract available. PMID 25470713
- [Result] Platzbecker U, Avvisati G, Cicconi L, Thiede C, Paoloni F, Vignetti M, Ferrara F, Divona M, Albano F, Efficace F, Fazi P, Sborgia M, Di Bona E, Breccia M, Borlenghi E, Cairoli R, Rambaldi A, Melillo L, La Nasa G, Fiedler W, Brossart P, Hertenstein B, Salih HR, Wattad M, Lubbert M, Brandts CH, Hanel M, Rollig C, Schmitz N, Link H, Frairia C, Pogliani EM, Fozza C, D'Arco AM, Di Renzo N, Cortelezzi A, Fabbiano F, Dohner K, Ganser A, Dohner H, Amadori S, Mandelli F, Ehninger G, Schlenk RF, Lo-Coco F. Improved Outcomes With Retinoic Acid and Arsenic Trioxide Compared With Retinoic Acid and Chemotherapy in Non-High-Risk Acute Promyelocytic Leukemia: Final Results of the Randomized Italian-German APL0406 Trial. J Clin Oncol. 2017 Feb 20;35(6):605-612. doi: 10.1200/JCO.2016.67.1982. Epub 2016 Oct 31. PMID 27400939
- [Derived] Chen S, Qin W, Lu X, Liu L, Zheng Y, Lu X, Wang X, Zhang X, Gong S, Wei S, Zhang H, Ding H, Seifollah R, Li J, Zhang H, Wu D, Abiona O, He P, Zhang R, Wald D, Wang H. Arsenic trioxide versus Realgar-Indigo naturalis formula in non-high-risk acute promyelocytic leukemia: a multicenter, randomized trial. Haematologica. 2025 Mar 1;110(3):621-628. doi: 10.3324/haematol.2024.285905. PMID 39506905
- [Derived] Zhang X, Liu L, Yao Y, Gong S, Wang M, Xi J, Chen L, Wei S, Zhang H, Zhao C, Wang H. Treatment of non-high-risk acute promyelocytic leukemia with realgar-indigo naturalis formula (RIF) and all-trans retinoid acid (ATRA): study protocol for a randomized controlled trial. Trials. 2020 Jan 2;21(1):7. doi: 10.1186/s13063-019-3983-2. PMID 31898521